CLINICAL TRIAL: NCT02707952
Title: A Randomized, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Japanese Adults With Chronic Hepatitis C Virus Infection (CERTAIN-1)
Brief Title: A Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Japanese Adults With Chronic Hepatitis C Virus Infection
Acronym: CERTAIN-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-594
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C Virus; Hepatitis C Virus
Keywords: Compensated cirrhosis; Non-cirrhotic; Renal impairment; Hepatitis C virus (HCV); Hepatitis C; Chronic Hepatitis C; Hepatitis C Genotype 1; Hepatitis C Genotype 2; Hepatitis C Genotype 3; Hepatitis C Genotype 4; Hepatitis C Genotype 5; Hepatitis C Genotype 6; DAA-experienced
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Renal Insufficiency | interventions — glecaprevir and pibrentasvir; glecaprevir; pibrentasvir; ombitasvir; paritaprevir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) once daily (QD) for 8 weeks in HCV genotype(GT)1 -infected, DAA treatment-naïve participants without cirrhosis.
  Interventions: Drug: ABT-493/ABT-530
- Arm B (Active Comparator): Ombitasvir (25 mg)/paritaprevir (150 mg)/ritonavir (100mg) (OBV/PTV/r) QD for 12 weeks in HCV GT1 infected, DAA treatment-naïve participants without cirrhosis.
  Interventions: Drug: OBV/PTV/r
- Arm C (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120mg) QD for 12 weeks in HCV GT1- or GT2-infected participants with compensated cirrhosis, HCV GT3-, 4-, 5- and 6-infected participants (with compensated cirrhosis or without cirrhosis), HCV GT1- and GT2-infected participants who had failed prior DAA treatments (with compensated cirrhosis or without cirrhosis), and HCV GT1- or GT2-infected participants with severe renal impairment and compensated cirrhosis.
  Interventions: Drug: ABT-493/ABT-530
- Arm D (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 8 weeks in GT1- or GT2-infected participants with severe renal impairment and without cirrhosis.
  Interventions: Drug: ABT-493/ABT-530

INTERVENTIONS:
Drug: ABT-493/ABT-530 — Co-formulated tablet
  Other Names: Glecaprevir/Pibrentasvir; glecaprevir (ABT-493); pibrentasvir (ABT-530)
  Arms: Arm A; Arm C; Arm D
Drug: OBV/PTV/r — Co-formulated tablet
  Other Names: Ombitasvir/paritaprevir/ritonavir; ombitasvir (ABT-267); paritaprevir (ABT-450); norvir (ritonavir)
  Arms: Arm B

SUMMARY:
The purpose of this phase 3, multicenter study is to evaluate the efficacy and safety of ABT-493/ABT-530 in Japanese adults with chronic Hepatitis C Virus (HCV)-infected, HCV direct-acting antiviral agent (DAA) treatment-naïve, and DAA treatment-experienced Japanese adult subjects.

DETAILED DESCRIPTION:
The study consisted of two sub-studies that enrolled in parallel. Substudy 1 was randomized, open-label, and active-controlled, wherein HCV treatment-naïve or interferon (IFN)-experienced (i.e., DAA treatment-naïve), genotype (GT)1-infected participants without cirrhosis were enrolled. Substudy 2 was non-randomized, open label, and enrolled special populations of HCV-infected participants [GT1- or GT2-infected subjects with compensated cirrhosis, HCV GT3-, 4-, 5- and 6-infected subjects (with compensated cirrhosis or without cirrhosis), HCV GT1- and GT2-infected subjects who had failed prior DAA treatments (with compensated cirrhosis or without cirrhosis), HCV GT1- or GT2-infected subjects with severe renal impairment (with compensated cirrhosis or without cirrhosis)].

ELIGIBILITY:
Inclusion Criteria:

* Females were postmenopausal for at least 2 years; surgically sterile or had a vasectomized partner; or, if of childbearing potential and sexually active with a male partner, were currently using at least 1 effective method of birth control at the time of Screening and agreed to practice 1 effective method of birth control from Screening through 30 days after stopping study drug. Sexually active males were surgically sterile or, if sexually active with a female partner of childbearing potential, agreed to practice 1 effective form of birth control from Screening through 30 days after stopping study drug.
* Screening central laboratory result indicated HCV single genotype infection for the appropriate treatment arm, without co-infection of any other genotype.
* Chronic HCV infection is defined as one of the following:

  * Positive for anti-HCV antibody (Ab) and/or HCV RNA at least 6 months before Screening.
  * A liver biopsy consistent with chronic HCV infection.
* Agreed to voluntarily sign and date an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) prior to the initiation of any screening or study specific procedures.
* Participants who were able to understand and adhere to the study visit schedule and all other protocol requirements.
* Absence of hepatocellular carcinoma (HCC) as indicated by an ultrasound, computed tomography (CT) scan or magnetic resonance imaging (MRI).

Exclusion Criteria:

* Females who were pregnant or planned to become pregnant, or breastfeeding or males whose partner was pregnant or planning to become pregnant during the study.
* Participants co-infected with hepatitis B virus or human immunodeficiency virus.
* Use of contraindicated medications or supplements within 2 weeks or 10 half-lives (if known), whichever was longer, prior to the first dose of any study drug.
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
* Any cause of liver disease other than chronic HCV infection.
* Any current or past clinical evidence of Child-Pugh B or C classification or clinical history of decompensated liver disease.
* Consideration by the investigator, for any reason, that the participant is an unsuitable candidate to receive ABT-493/ABT-530.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2017-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

REFERENCES:
- [Background] Chayama K, Suzuki F, Karino Y, Kawakami Y, Sato K, Atarashi T, Naganuma A, Watanabe T, Eguchi Y, Yoshiji H, Seike M, Takei Y, Kato K, Alves K, Burroughs M, Redman R, Pugatch DL, Pilot-Matias TJ, Krishnan P, Oberoi RK, Xie W, Kumada H. Efficacy and safety of glecaprevir/pibrentasvir in Japanese patients with chronic genotype 1 hepatitis C virus infection with and without cirrhosis. J Gastroenterol. 2018 Apr;53(4):557-565. doi: 10.1007/s00535-017-1391-5. Epub 2017 Sep 25. PMID 28948366
- [Derived] Brown RS Jr, Collins MA, Strasser SI, Emmett A, Topp AS, Burroughs M, Ferreira R, Feld JJ. Efficacy and Safety of 8- or 12 Weeks of Glecaprevir/Pibrentasvir in Patients with Evidence of Portal Hypertension. Infect Dis Ther. 2022 Apr;11(2):913-924. doi: 10.1007/s40121-022-00599-8. Epub 2022 Feb 17. PMID 35174470
- [Derived] Naganuma A, Chayama K, Notsumata K, Gane E, Foster GR, Wyles D, Kwo P, Crown E, Bhagat A, Mensa FJ, Otani T, Larsen L, Burroughs M, Kumada H. Integrated analysis of 8-week glecaprevir/pibrentasvir in Japanese and overseas patients without cirrhosis and with hepatitis C virus genotype 1 or 2 infection. J Gastroenterol. 2019 Aug;54(8):752-761. doi: 10.1007/s00535-019-01569-7. Epub 2019 Mar 13. PMID 30868245
- [Derived] Krishnan P, Schnell G, Tripathi R, Beyer J, Reisch T, Dekhtyar T, Irvin M, Xie W, Fu B, Burroughs M, Redman R, Kumada H, Chayama K, Collins C, Pilot-Matias T. Integrated Resistance Analysis of CERTAIN-1 and CERTAIN-2 Studies in Hepatitis C Virus-Infected Patients Receiving Glecaprevir and Pibrentasvir in Japan. Antimicrob Agents Chemother. 2018 Jan 25;62(2):e02217-17. doi: 10.1128/AAC.02217-17. Print 2018 Feb. PMID 29180522
- [Derived] Yartel AK, Rein DB, Brown KA, Krauskopf K, Massoud OI, Jordan C, Kil N, Federman AD, Nerenz DR, Brady JE, Kruger DL, Smith BD. Hepatitis C virus testing for case identification in persons born during 1945-1965: Results from three randomized controlled trials. Hepatology. 2018 Feb;67(2):524-533. doi: 10.1002/hep.29548. Epub 2018 Jan 2. PMID 28941361
- [Derived] Toyoda H, Chayama K, Suzuki F, Sato K, Atarashi T, Watanabe T, Atsukawa M, Naganuma A, Notsumata K, Osaki Y, Nakamuta M, Takaguchi K, Saito S, Kato K, Pugatch D, Burroughs M, Redman R, Alves K, Pilot-Matias TJ, Oberoi RK, Fu B, Kumada H. Efficacy and safety of glecaprevir/pibrentasvir in Japanese patients with chronic genotype 2 hepatitis C virus infection. Hepatology. 2018 Feb;67(2):505-513. doi: 10.1002/hep.29510. Epub 2017 Nov 24. PMID 28865152
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-treat population: all participants who received at least 1 dose of study drug
Groups:
- Arm A: ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) once daily (QD) for 8 weeks in HCV genotype 1 (GT1) -infected, DAA treatment-naïve participants without cirrhosis.
- Arm C: ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 12 weeks in HCV GT1- or GT2-infected participants with compensated cirrhosis, HCV GT3-, 4-, 5- and 6-infected participants (with compensated cirrhosis or without cirrhosis), HCV GT1- and GT2-infected participants who had failed prior DAA treatments (with compensated cirrhosis or without cirrhosis), and HCV GT1- or GT2-infected participants with severe renal impairment and compensated cirrhosis.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started (This milestone represents participants randomized.) | 129 | 53 | 103 | 10
Participants Who Received Study Drug | 129 | 52 | 103 | 10
Completed | 127 | 52 | 101 | 10
Not Completed | 2 | 1 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug (ITT population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Total
Number analyzed (Participants) | 129 | 52 | 103 | 10 | 294
Age, Customized [Number; unit: participants]
  < 65 years | 66 | 22 | 33 | 4 | 125
  >= 65 years to < 75 years | 37 | 23 | 43 | 4 | 107
  >= 75 years | 26 | 7 | 27 | 2 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 38 | 58 | 6 | 184
  Male | 47 | 14 | 45 | 4 | 110

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Arms A and B With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants who received at least 1 dose of study drug, excluding participants with the Y93H polymorphism in NS5A at baseline (ITT-PS population); participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 106 | 52
percentage of participants | 99.1 | 100
Statistical Analysis 1: Comparison: Arm A vs Arm B; Test type: Non-Inferiority — The percentage of participants achieving SVR12 was calculated for each arm and a 2-sided 95% CI for the difference in SVR12 rates (Arm A minus Arm B) was calculated using the normal approximation to the binomial distribution to assess non-inferiority in SVR12 rates of arm A to arm B. If the lower bound of the confidence interval (CI) for the difference was above the non-inferiority margin of -10%, then arm A was considered non-inferior to arm B; Rate Difference = -0.9, 95% CI 2-sided [-2.8 to 0.9] — 95% CI was calculated using the normal approximation to the binomial distribution

2. Secondary Outcome: Percentage of Participants in Arm A With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. 95% CI was calculated using the normal approximation to the binomial distribution.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat (ITT) population: all participants who received at least 1 dose of study drug; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A
Number analyzed (Participants) | 129
percentage of participants | 99.2 [97.7 to 100.0]

3. Secondary Outcome: Percentage of Participants for Each Sub-Population in Arms C and D With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. Subpopulations defined as Genotype 1 and 2 infected cirrhotic participants, prior direct acting antiviral agent (DAA) treatment experienced (T-exp) participants, Genotype 3, 4, 5 or 6-infected participants, and participants with severe renal impairment (RI). 95% CI was calculated using the Wilson score method.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population); participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm C | Arm D
Number analyzed (Participants) | 103 | 10
percentage of participants
  HCV GT1 Participants with Compensated Cirrhosis: number analyzed (Participants) | 38 | 0
  HCV GT1 Participants with Compensated Cirrhosis | 100 [90.8 to 100.0] |
  HCV GT2 Participants with Compensated Cirrhosis: number analyzed (Participants) | 18 | 0
  HCV GT2 Participants with Compensated Cirrhosis | 100 [82.4 to 100.0] |
  DAA Experienced Participants: number analyzed (Participants) | 33 | 0
  DAA Experienced Participants | 93.9 [80.4 to 98.3] |
  HCV GT3,4,5 and 6 Participants: number analyzed (Participants) | 12 | 0
  HCV GT3,4,5 and 6 Participants | 83.3 [55.2 to 95.3] |
  Participants With Severe RI and with Cirrhosis: number analyzed (Participants) | 2 | 0
  Participants With Severe RI and with Cirrhosis | 100.0 [34.2 to 100.0] |
  Participants With Severe RI and without Cirrhosis: number analyzed (Participants) | 0 | 10
  Participants With Severe RI and without Cirrhosis |  | 100 [72.2 to 100.0]

4. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline HCV RNA during treatment; confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment, or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment. 95% CI was calculated using the Wilson score method.
Time Frame: Treatment Weeks 1, 2, 4, 8 (end of treatment for 8-week treatment arm), and 12 (end of treatment for 12-week treatment arm) or premature discontinuation from treatment
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 129 | 52 | 103 | 10
percentage of participants | 0 [0.0 to 2.9] | 0 [0.0 to 6.9] | 1.0 [0.2 to 5.3] | 0 [0.0 to 27.8]

5. Secondary Outcome: Percentage of Participants With Post-Treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants with HCV RNA levels < LLOQ at the end of treatment, excluding participants who were been shown to be re-infected. The confidence interval was calculated using the Wilson score method.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population) with at least one post-treatment HCV RNA value, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 129 | 51 | 100 | 10
percentage of participants | 0 [0.0 to 2.9] | 0 [0.0 to 7.0] | 3.0 [1.0 to 8.5] | 0 [0.0 to 27.8]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16 weeks). Serious adverse events (SAEs) were collected starting from the time that the informed consent was signed until the end of the study (up to 21 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) or serious adverse event (SAE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ARM A | ARM B | ARM C | ARM D
Serious Adverse Events (participants affected / at risk) | 0/129 | 3/52 | 0/103 | 1/10
Other Adverse Events (participants affected / at risk) | 51/129 | 28/52 | 44/103 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=129) | ARM B (N=52) | ARM C (N=103) | ARM D (N=10)
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=129) | ARM B (N=52) | ARM C (N=103) | ARM D (N=10)
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
EYE PRURITUS (Eye disorders) | 0 | 0 | 0 | 1
GINGIVAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 4 | 1 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 3 | 1
MALAISE (General disorders) | 3 | 0 | 6 | 0
PYREXIA (General disorders) | 0 | 3 | 2 | 1
CYSTITIS (Infections and infestations) | 1 | 3 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 20 | 7 | 9 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 3 | 3 | 4 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 2
BLOOD MAGNESIUM INCREASED (Investigations) | 0 | 0 | 0 | 1
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 0 | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 2 | 1
PROTEIN URINE PRESENT (Investigations) | 1 | 1 | 0 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
HEADACHE (Nervous system disorders) | 6 | 5 | 7 | 1
INSOMNIA (Psychiatric disorders) | 1 | 0 | 0 | 1
RENAL DISORDER (Renal and urinary disorders) | 0 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 8 | 5 | 13 | 0
RASH (Skin and subcutaneous tissue disorders) | 3 | 3 | 6 | 1
HYPERTENSION (Vascular disorders) | 4 | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.